CLINICAL TRIAL: NCT00289653
Title: Smoking While on Transdermal Nicotine Replacement Therapy: Effects on Craving and Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Dr. Peter Selby, Dr. P. Selby, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205/2005
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2017-12

CONDITIONS: Nicotine Dependence
Keywords: nicotine dependence,; transdermal nicotine patch,; smoking while receiving nicotine replacement,; comorbidities
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single open-label treatment arm (Experimental): Adult smokers willing to quit were treated with escalating doses of transdermal nicotine patch (Nicoderm) and brief counselling if they continued to smoke over a 9-week treatment period.
  Interventions: Drug: Nicoderm

INTERVENTIONS:
Drug: Nicoderm
  Other Names: NRT patch; nicotine patch

SUMMARY:
Smoking while on nicotine patches will help subjects to reduce their expired carbon monoxide levels from the levels they were before they started using the patch. Subjects will also decrease their daily consumption of cigarettes.

DETAILED DESCRIPTION:
Subjects who smoke while on an individually dosed tNRT will reduce their expired carbon monoxide levels from pre- to post-treatment conditions. They will also decrease their daily consumption of cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* at least 19 years of age
* male or female
* have intention to quit smoking within the next 6 months
* smoke 10 or more cigarettes per day

Exclusion Criteria:

* Pregnant or not using an adequate enough method of birth control to ensure that they are not at risk of becoming pregnant
* breastfeeding
* have any generalized skin disorders
* are in an immediate post-myocardial infarction period or have life-threatening arrhythmias, have severe or worsening angina pectoris or have had a recent cerebral vascular accident
* are using additional nicotine replacement therapies or any other smoking cessation pharmacotherapy
* any clinically significant ECG abnormalities
* any known hypersensitivity to components of the transdermal system

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter L. Selby, MBBS, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Selby P, Andriash K, Zawertailo L, Persad D, Zack M, Busto UE. Escalating doses of transdermal nicotine in heavy smokers: effects on smoking behavior and craving. J Clin Psychopharmacol. 2013 Oct;33(5):667-74. doi: 10.1097/JCP.0b013e31829a829d. PMID 23963055

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine Therapy + Counselling: Nicotine replacement therapy + brief counselling
Period: Overall Study
Arm/Group | Nicotine Therapy + Counselling
Started | 23
Completed | 12
Not Completed | 11

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Participants: All eligible enrolled participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Mean Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 25.7 (13.4)
Carbon monoxide gas (CO) reading [Mean (Standard Deviation); unit: ppm] | 23.1 (11.5)
No. of previous serious quit attempts [Mean (Standard Deviation); unit: Quit attempts] | 4.7 (6.3)
No. years smoking [Mean (Standard Deviation); unit: years] | 30.1 (12.9)
Fagerstrom Test of Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — A standard test to assess nicotine dependence completed by the subject. The yes/ no responses are scored 0-1 and multiple choice answers are scored 0-3.
  Items are summed to yield a total score of 0-10. Total score indicates level of nicotine dependence. 0-2 (Low); 3-5 (Low-moderate); 5-7 (Moderate); 8-10 (High).
  units on a scale | 6.3 (2.3)
Hamilton Depression Rating Scale (HAM-D) [Mean (Standard Deviation); unit: units on a scale] — This measure is used to assess level of depression. There are 21 items and the score is based on the first 17 items. 8 items are scored 0-4. 9 items are scored 0-2. Total score determines level of depression. 0-7 (normal); 8-13 (mild depression); 14-18 (moderate depression); 19-22 (severe depression); => 23 (very severe depression)
  units on a scale | 8.9 (9.8)
Beck Depression Inventory (BDI) score [Mean (Standard Deviation); unit: units on a scale] — This self report scale measures level of depression. the response of each of the 21 items ranges from 0-3. The total score (range 0-63) reflects level of depression. 0-10 (normal) 11-16 (moderate) 17-20 (borderline) 21-30 (moderate) 21-40 (Severe) > 40 (extreme)
  units on a scale | 10.0 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: Carbon Monoxide Levels
Description: Expired Co levels were measured to confirm smoking status
Time Frame: measured at week 10
Measure: Mean (Standard Deviation); unit: parts per million
Groups:
- Enrolled Participants: 12 participants who completed the study
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 12
parts per million | 9.2 (6.3)

2. Secondary Outcome: Smoking Cessation
Description: self reported # cigarettes per day
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: cigarettes per day
Groups:
- Enrolled Participants: participants who completed the study
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 12
cigarettes per day | 3.7 (4.0)

ADVERSE EVENTS:
Time Frame: 10 weeks
Groups:
- Enrolled Participants: participants who enrolled in the study
Arm/Group | Enrolled Participants
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 17/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Participants (N=23)
adverse event- respiratory infection and colds (Respiratory, thoracic and mediastinal disorders) | 6 (9) — Adverse event (non-serious) unrelated to NRT
Skin irritation (Product Issues) | 8 (8) — Reaction to Nicotine patch -Skin irritation
sleep disturbance (Product Issues) | 7 (8) — reaction to nicotine patch
Nausea and Vomitting (Product Issues) | 5 (5) — Reaction to nicotine patch
Emotional Distress (Social circumstances) | 2 (2)
Depressive Symptoms (Psychiatric disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No